CLINICAL TRIAL: NCT01064739
Title: Renal Salt Handling in Postural Tachycardia Syndrome Following Dietary Dopa Administration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Emily M. Garland, Research Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PN 1767
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Participants
Keywords: Healthy Volunteers; Fava bean consumption; L-Dopa content in Fava Beans; Sodium; Potassium; Electrolyte Balance; Natriuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Diet +/- fava beans (Experimental): Participants underwent testing while on a methylxanthine-free diet providing 150 mEq sodium and 75 mEq potassium per day. The study involved a longitudinal design where the participants served as their own controls. Subjects consumed the standard fixed sodium diet on study day one. On study day two, participants ate 100 g of puréed fava beans and pods with study diet at breakfast (0800hr) and lunch (1200hr).
  Interventions: Dietary Supplement: Fava beans; Other: Fixed Sodium Diet

INTERVENTIONS:
Dietary Supplement: Fava beans — Participants will receive 100g of fresh fava beans for breakfast and lunch on one study day and prior to this study day will be restricted to a fixed sodium low monoamine diet
Other: Fixed Sodium Diet — Fixed sodium low monoamine diet

SUMMARY:
The purpose of this study is to learn how plants can play a role in gain/loss of sodium in the urine and in the regulation of blood pressure. Dopamine is a chemical mostly present in the brain and kidneys which assists in regulation of the body's salts (sodium and potassium). Fava beans contain a lot of the chemical that increases the production of dopamine by the kidneys.

The purpose of these studies is to characterize the diuretic effects of dietary catecholamine sources in healthy individuals. Specific aims are:

1. To determine the effect of dietary dopa sources on plasma and urinary catecholamines.
2. To investigate the capacity of botanical dopaminergic agents (fava beans) to induce natriuresis in a short term study.
3. To provide preliminary data on the effects of dietary dopa on heart rate and blood pressure.

In these studies, we will test the null hypothesis (Ho) that urinary sodium excretion will not differ in healthy volunteers after consumption of a fixed-sodium study diet and the study diet plus fava beans.

DETAILED DESCRIPTION:
Fava beans are a broad bean, with potential clinical relevance in Parkinson's patients since they contain high levels of the dopamine precursor, dihydroxyphenylalanine (dopa).In addition to the central nervous system functions of dopamine that are compromised in Parkinson's disease, renal dopamine has vasodilatory and natriuretic activity. Elevated urinary dopamine, however, does not consistently correlate with increased urinary sodium excretion, and there are conflicting opinions over the conditions under which renal dopamine might regulate sodium balance.The goal of our study was to clarify the natriuretic effect of fava beans, obtained from a source that serves patients with Parkinson's disease. Catechol and sodium data were compared in healthy volunteers using a longitudinal design in which all participants consumed a fixed sodium study diet on day 1 and the fixed sodium diet plus fava beans on day 2. Blood was sampled at 1, 2, 4 and 6 hours after breakfast, and three consecutive 4-hr urine samples were collected.

Postural tachycardia syndrome (POTS) is the most common form of orthostatic intolerance, affecting an estimated 500,000 Americans, principally young women. POTS refers to an excessive increase in heart rate (>30 beats per minute) on standing in the absence of orthostatic hypotension. Previous findings by the Robertson/Garland research group suggest that mechanisms involved in orthostatic and absolute volume regulation contribute to POTS pathophysiology. A follow-up study might compare the influences of diet in patients with POTS and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Free of medications with the potential to influence BP
* Age between 18-60 years
* Male and female subjects are eligible
* Able and willing to provide informed consent

Exclusion Criteria:

* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or screening results
* Positive urine b-hcg pregnancy test
* Evidence of cardiac structural disease (by clinical examination or prior echocardiogram)
* Hypertension defined as a BP>145/95 (off medications) or need for antihypertensive medications
* Evidence of significant conduction system delay (QRS duration >120 ms) on electrocardiogram
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol Food allergies to favas or other dietary dopa sources selected
* Parkinson's Disease
* Diagnosis of Glucose-6-Phosphate Dehydrogenase (G6P) Deficiency or Individuals from the Mediterranean with family history of G6PD.
* Prolonged QT interval on ECG> 480 13. Familial history of sudden cardiac death

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Garland, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garland EM, Cesar TS, Lonce S, Ferguson MC, Robertson D. An increase in renal dopamine does not stimulate natriuresis after fava bean ingestion. Am J Clin Nutr. 2013 May;97(5):1144-50. doi: 10.3945/ajcn.112.048470. Epub 2013 Apr 3. PMID 23553159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the Nashville, TN area between November, 2009 and November, 2010.
Groups:
- Fixed Sodium Diet +/- Fava Beans: Participants consumed a fixed sodium diet on day 1 and the same diet plus 100g of fresh fava beans at breakfast and lunch on day 2.The 14 participants received both interventions.
Period: Fixed Sodium Study Diet
Arm/Group | Fixed Sodium Diet +/- Fava Beans
Started | 14 (14 participants consumed the fixed-sodium study diet prior to the fava bean supplement study day.)
Completed | 14
Not Completed | 0
Period: Fixed Sodium Diet + Fava Beans
Arm/Group | Fixed Sodium Diet +/- Fava Beans
Started | 14
Completed | 13 (1 participant withdrew with blood in his urine on the fava bean study day.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Fava Beans: A meal enriched in dopa content, using fava beans, will be eaten at 0800hr (breakfast) and 1200hr (lunch), with measurements following the same schedule as the day with just fixed sodium study diet.
  Fava beans : Participants will receive 100g of fresh fava beans for breakfast and lunch on one study day and prior to this study day will be restricted to a fixed sodium low monoamine diet
Arm/Group | Fava Beans
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Plasma Dopa 1 hr After Breakfast
Description: Subjects consumed the standard fixed sodium diet for at least two days prior to study and on study day one during an inpatient stay in the Vanderbilt Clinical Research Center. On study day two, participants ate 100 g of puréed fava beans and pods with study diet at breakfast (0800hr) and lunch (1200hr). Blood was sampled for catechol assays before and at 1, 2, 4 and 6 hours after breakfast. Plasma dopa 1 hour after breakfast was specified as a primary outcome. Other catechols (dihydroxyphenylglycol, norepinephrine, epinephrine, dopamine, dihydroxyphenylacetic acid) and other time points (2, 3, 4, 6hr after breakfast) are non-primary outcomes.
Time Frame: Plasma samples collected 1 hour after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Fixed Sodium Study Diet: A study diet with a fixed amount of sodium and no fava beans.
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
pg/mL | 11670 (5440) | 1705 (530)

2. Secondary Outcome: Plasma Dopa 2 Hrs After Breakfast
Description: as for outcome 1
Time Frame: Plasma samples collected 2 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Fixed Sodium Study Diet: Participants underwent testing while on a methylxanthine-free diet providing 150 mEq sodium and 75 mEq potassium per day. The study involved a longitudinal design where the participants served as their own controls. Subjects consumed the standard fixed sodium diet on study day one. On study day two, participants ate 100 g of puréed fava beans and pods with study diet at breakfast (0800hr) and lunch (1200hr).
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 1689 (451) | 8122 (3626)

3. Secondary Outcome: Plasma Dopa 4 Hrs After Breakfast
Description: as for outcome 1
Time Frame: Plasma samples collected 4 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 12 | 12
pg/mL | 1800 (608) | 3473 (1106)

4. Primary Outcome: Urinary Dopa
Description: Urinary dopa excreted 4-8 hours after breakfast was specified as a primary outcome. Other catechols (dihydroxyphenylglycol, norepinephrine, epinephrine, dopamine, dihydroxyphenylacetic acid) and other time points (0-4 hr, 8-12 hr after breakfast) are non-primary outcomes.
Time Frame: 4-8 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Groups:
- Fixed Sodium Study Diet: Participants underwent testing while on a methylxanthine-free diet providing 150 mEq sodium and 75 mEq potassium per day. The study involved a longitudinal design where the participants served as their own controls. Subjects consumed the standard fixed sodium diet on study day. On study day two, participants ate 100 g of puréed fava beans and pods with study diet at breakfast (0800hr) and lunch (1200hr).
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
micrograms/4hr | 24.2 (21.2) | 4.4 (3.0)

5. Primary Outcome: Urinary Sodium
Description: Urinary sodium excreted 4-8 hours after breakfast was designated as a primary outcome. Other urine samples (0-4 hr, 8-12 hr after breakfast) are considered as non-primary outcomes.
Time Frame: 4 to 8 hours after breakfast
Measure: Mean (Standard Deviation); unit: mEq/4 hr
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
mEq/4 hr | 24 (8.8) | 35 (17)

6. Secondary Outcome: Plasma Dopa 6 Hrs After Breakfast
Description: as for outcome 1
Time Frame: Plasma samples collected 6 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 1712 (488) | 7385 (3489)

7. Secondary Outcome: Plasma Norepinephrine
Description: Plasma norepinephrine 1 hour after breakfast
Time Frame: 1 hour after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 188 (72) | 228 (132)

8. Secondary Outcome: Plasma Norepinephrine
Description: Plasma norepinephrine 2 hours after breakfast
Time Frame: 2 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 173 (114) | 304 (226)

9. Secondary Outcome: Plasma Norepinephrine
Description: Plasma norepinephrine 4 hours after breakfast
Time Frame: 4 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 12 | 12
pg/mL | 155 (74) | 266 (220)

10. Secondary Outcome: Plasma Norepinephrine
Description: Plasma norepinephrine 6 hours after breakfast
Time Frame: 6 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
pg/mL | 354 (273) | 159 (89)

11. Secondary Outcome: Plasma Dopamine
Description: Plasma dopamine 1 hour after breakfast
Time Frame: 1 hour after breakfast
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
pg/mL | 90 (47) | 6 (3)

12. Secondary Outcome: Plasma Dopamine
Description: Plasma dopamine 2 hours after breakfast
Time Frame: 2 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 7.4 (2.9) | 93.8 (54.1)

13. Secondary Outcome: Plasma Dopamine
Description: Plasma dopamine 4 hours after breakfast
Time Frame: 4 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 12 | 12
pg/mL | 6.7 (2.8) | 50.3 (26.6)

14. Secondary Outcome: Plasma Dopamine
Description: Plasma dopamine 6 hours after breakfast
Time Frame: Plasma samplesPlasma dopamine 6 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
pg/mL | 7.9 (3.1) | 91.3 (41.9)

15. Secondary Outcome: Urinary Dopa
Description: Urinary dopa excreted 4-8 hours after breakfast was specified as a primary outcome. Other time points (0-4 hr, 8-12 hr after breakfast) are non-primary outcomes.
Time Frame: 0-4 hours after breakfast
Measure: Mean (Standard Deviation); unit: ug/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 10 | 10
ug/4hr | 3.80 (2.13) | 22.09 (13.42)

16. Secondary Outcome: Urinary Dopa
Description: as for outcome 15
Time Frame: 8-12 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
micrograms/4hr | 3.43 (1.31) | 5.43 (2.78)

17. Secondary Outcome: Urinary Dopamine
Description: Urinary dopamine excreted 0 to 4 hours after breakfast
Time Frame: 0 to 4 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 10 | 10
micrograms/4hr | 45.3 (21.4) | 306.3 (116.2)

18. Secondary Outcome: Urinary Dopamine
Description: Urinary dopamine excreted 4 to 8 hours after breakfast
Time Frame: 4 to 8 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4 hours
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
micrograms/4 hours | 360 (235) | 54.0 (29.5)

19. Secondary Outcome: Urinary Dopamine
Description: Urinary dopamine excreted 8 to 12 hours after breakfast
Time Frame: 8 to 12 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
micrograms/4hr | 44.2 (17.0) | 159.2 (111.5)

20. Secondary Outcome: Urinary Norepinephrine
Description: Urinary norepinephrine excreted 0-4 hours after breakfast
Time Frame: 0 to 4 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4 hours
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
micrograms/4 hours | 11.7 (5.1) | 5.1 (2.3)

21. Secondary Outcome: Urinary Norepinephrine
Description: Urinary norepinephrine excreted 4-8 hours after breakfast
Time Frame: 4 to 8 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
micrograms/4hr | 8.43 (6.25) | 13.26 (6.99)

22. Secondary Outcome: Urinary Norepinephrine
Description: Urinary norepinephrine excreted 8-12 hours after breakfast
Time Frame: 8 to 12 hours after breakfast
Measure: Mean (Standard Deviation); unit: micrograms/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
micrograms/4hr | 6.72 (6.77) | 11.35 (3.44)

23. Secondary Outcome: Supine Systolic Blood Pressure
Description: Supine systolic blood pressure 6 hours after breakfast
Time Frame: Supine-6 hours after breakfast on both study days.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
mm Hg | 104 (7) | 102 (8)

24. Secondary Outcome: Supine Heart Rate
Description: Supine heart rate 6 hours after breakfast
Time Frame: 6 hours after breakfast
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Number analyzed (Participants) | 13 | 13
beats per minute | 66 (13) | 65 (15)

25. Secondary Outcome: Urinary Sodium
Description: Urinary sodium excreted 0-4 hours after breakfast.
Time Frame: 0-4 hours after breakfast
Measure: Mean (Standard Deviation); unit: mEq/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 10 | 10
mEq/4hr | 29.9 (11.4) | 23.5 (6.5)

26. Secondary Outcome: Urinary Sodium
Description: urinary sodium 8-12 hours after breakfast
Time Frame: 8-12 hours after breakfast
Measure: Mean (Standard Deviation); unit: mEq/4hr
Arm/Group | Fixed Sodium Study Diet | Fava Beans
Number analyzed (Participants) | 13 | 13
mEq/4hr | 32.5 (17.3) | 14.5 (6.9)

ADVERSE EVENTS:
Time Frame: 2 1/2 years
Arm/Group | Fava Beans | Fixed Sodium Study Diet
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fava Beans (N=14) | Fixed Sodium Study Diet (N=14)
blood in urine (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes